CLINICAL TRIAL: NCT02804906
Title: Rehabilitation in the Home Setting for Older Adults In the Early Period After Myocardial Infarction
Acronym: RESILIENT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 16-00554
Record Dates: First submitted 2016-06-14; First posted 2016-06-17 (Estimated); Last update posted 2020-01-22 (Actual); Status verified 2020-01

CONDITIONS: Acute Myocardial Infarction (AMI)

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Home-Based Physical Therapy (Experimental)
  Interventions: Behavioral: Home-based physical therapy
- Control-30-minute counseling session (Active Comparator): Participants in the control arm will be provided with a 30-minute counseling session on risk factor modification prior to discharge.
  Interventions: Behavioral: Usual Care

INTERVENTIONS:
Behavioral: Home-based physical therapy — Participants will be visited by a physical therapist 3 times a week for approximately 1 hour each day, for a duration of 4 weeks. These visits will serve to encourage adherence to the intervention, reinforce activities recommended at discharge, monitor safety under direct supervision, and adjust the exercise prescription if/as needed (e.g. advance recommended activity level) if necessary. Patients will also be provided with a tablet computer device installed with software, Moving Analytics, that will reinforce the cardiac rehabilitation program through daily reminders and easily accessible visual activity plans. This program will be updated by the physical therapist during home visits as the program advances. Daily patient-reported health status ("Your Activities of Daily Living") 26 will be ascertained on the same tablet device by participants three times per week using open source software designed.
  Arms: Home-Based Physical Therapy
Behavioral: Usual Care — Participants in the control arm will be provided with a 30-minute counseling session on risk factor modification prior to discharge. Participants will be provided with a tablet computer device to complete patient-reported health status ("Your Activities of Daily Living") 26 three times per week using open source software designed. Participants will be visited by the Research Coordinator or member of the study team at one month post-hospital discharge to perform a follow-up assessment that will include ADLs, IADLs, SF-12 PCS, frailty measures, and questions on healthcare utilization (hospital readmissions).
  Arms: Control-30-minute counseling session

SUMMARY:
This pilot feasibility study will test whether a home-based cardiac rehabilitation intervention, using physical therapist visits combined with mobile health technology, will prevent decline in high-risk patients post acute myocardial infarction (AMI). Participants will be randomized to either an intervention arm (home-based physical therapy), or a control (usual care) arm. Prior to discharge, participants in the intervention arm will receive a 1-hour educational session by a research physical therapist that includes information on cardiac risk factor management, postoperative recovery, education on medication adherence, and a prescription for home exercise that is tailored to each patient's baseline abilities and limitations. Participants assigned to the control arm will receive a 30-minute counseling session on risk factor modification prior to discharge, in addition to usual care post-AMI.

DETAILED DESCRIPTION:
All participants enrolled in this research study will receive the FDA-approved FitBit Flex, a wearable activity monitoring device which will objectively measure physical activity and sedentary behavior in the period post-hospital discharge. Daily activity monitoring will include: number of steps, distance traveled, calories burned, number of active minutes.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of acute myocardial infarction (AMI).

Exclusion Criteria:

* moderate to severe cognitive impairment; non-ambulatory
* severe heart failure (NYHA Class IV); decisional impairment as assessed by the University of California
* San Diego Brief Assessment of Capacity to Consent (UBACC) 22, if the RC questions capacity; very limited life expectancy (e.g. anticipated discharge to hospice)
* non-English/non-Spanish speaking.

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 27 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2018-12-14 (Actual); Study Completion 2019-01-14 (Actual)

PRIMARY OUTCOMES:
Activities of Daily Living (ADL) Decline | 5 Weeks
  Assessment of the functional dependence or independence in carrying out activities of daily living, including bathing, dressing, toileting, transferring, continence, and feeding.

SECONDARY OUTCOMES:
Decline in self-perceived physical health (measured by SF-12 PCS) | 5 Weeks
  Health status measure that addresses both physical and mental health.
Mean time spent in sedentary activity | 5 Weeks
Mortality Rate | 5 Weeks
Hospital readmission rate | 5 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: John Dodson, MD, Principal Investigator — New York University Medical School
Locations (1):
- New York University School of Medicine, New York, New York, United States